CLINICAL TRIAL: NCT03403803
Title: Prognosis and Therapeutic Biomarkers for Glioblastoma Patients
Status: Terminated | Type: Observational
Why Stopped: Were not able to meet enrollment goal due to inclusion/exclusion criteria
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 160280
Record Dates: First submitted 2017-11-09; First posted 2018-01-19 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Brain Tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva and CSF (cerebrospinal fluid)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Control Group
- Optune Only
  Interventions: Device: Optune
- Optune and TMZ
  Interventions: Device: Optune

INTERVENTIONS:
Device: Optune — Optune is a wearable and portable, FDA-approved device that has been shown in clinical trials to safely deliver continuous therapy to the area of your brain where your GBM (Glioblastoma) tumor is located.
  TMZ (Temozolomide) is an oral chemotherapy drug. It is an alkylating agent used as a treatment of some brain cancers; as a second-line treatment for astrocytoma and a first-line treatment for glioblastoma multiforme.
  Other Names: TMZ
  Groups: Optune Only; Optune and TMZ

SUMMARY:
The purpose of this study is to investigate if the potential biomarkers identified could be used for facilitating the diagnosis and prognosis of patients with glioblastoma (GBM).

DETAILED DESCRIPTION:
The objective of this proposed study is to determine the expression levels of a panel of markers including CD133, CD44, ABCC3, TNFRSF1A, AKT1, IDH2, and MGMT in GBM tissues and the CSF, blood, and saliva from patients with GBM receiving different types of treatment (Optune only or Optune with TMZ) and the non-brain tumor patients (controls). Our aims are: 1) To compare the differences of CD44 between the control group and the combined cancer groups at baseline; and 2) To compare the levels of CD44 and other markers among the 3 different groups such as control vs. GBM patients and Optune vs. Optune + TMZ after 8 weeks of treatment. Exploratory analysis of all other markers will be performed.

ELIGIBILITY:
Inclusion Criteria:

* 22 years old
* Control Group (only patients evaluated for neurological disorders whose evaluation require a lumbar puncture)
* Non-Control Group - Diagnosed with GBM (Glioblastoma)

Exclusion Criteria:

* Pregnancy
* Infectious Disease to include cold, flu, HIV, etc.
* Blood Disorder (example:low platelets, anemia, thrombosis)
* Vascular Malformations

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed with GBM or diagnosed with other neurological disorder that requires a lumbar puncture.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Primary Outcome - CD44 expression in cerebrospinal fluid (CSF), blood and saliva | 2 years
  Currently, Glioblastoma is only diagnosed and monitored with brain scans. Expression levels of CD44 along with CD133, ABCC3, TNFRSF1A, AKT1, IDH2 and MGMT in samples of CSF, blood and saliva from patients receiving different types of treatment and comparing them with non-GBM patients (control group) will be tested.

CONTACTS AND LOCATIONS:
Overall Officials: Ekokobe Fonkem, MD, Principal Investigator — Baylor Scott and White Medical Center, Temple, TX
Locations (1):
- Baylor Scott and White Medical Center, Temple, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT03403803/Prot_000.pdf
  • Informed Consent Form: Main Consent (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT03403803/ICF_001.pdf
  • Informed Consent Form: Control Consent (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT03403803/ICF_002.pdf